CLINICAL TRIAL: NCT02124967
Title: Exploring the Feasibility, Acceptability, and Effectiveness of a Mosque-Based Intervention to Promote Physical Activity in South Asian Muslim Women: A Pilot Study
Brief Title: A Mosque-Based Intervention to Promote Physical Activity in South Asian Muslim Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Jennifer Price, Advance Practice Nurse, Cardiology, Women's College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014-0029-B
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): A one hour exercise session which includes both aerobic activity and resistance training
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — A one hour exercise class including both aerobic activity and resistance training

SUMMARY:
South Asian (SA) women living in Ontario have a higher risk of developing type 2 diabetes and coronary heart disease (CHD) compared to the general population. Various explanations for these differences have been established, one of which is based on low levels of physical activity in people of SA origin, particularly in Muslim women.

This pilot trial will test the feasibility, acceptability and effectiveness of a Mosque-based exercise and educational intervention designed for SA Muslim women.

1. What is the feasibility of a mosque-based intervention to promote physical activity that is culturally and gender sensitive to South Asian Muslim women?
2. What is the acceptability of a mosque-based intervention to promote physical activity that is culturally and gender sensitive to South Asian Muslim women?
3. What is the effectiveness of a mosque-based intervention to promote physical activity that is culturally and gender sensitive to South Asian Muslim women?

DETAILED DESCRIPTION:
South Asian (SA) women (people with origins in Pakistan, India, Bangladesh or Sri Lanka) living in Ontario have a higher risk of developing type 2 diabetes and coronary heart disease (CHD) compared to the general population. Various explanations for these differences have been established, one of which is based on low levels of physical activity in people of SA origin, particularly in Muslim women. Studies suggest that they participate in less physical activity or recreational exercise compared to other SA women. Practical barriers (e.g. lack of time, childcare) are often interwoven with cultural barriers, such as restrictions leaving the home alone to enter mixed-gender settings, and lack of socialization into sporting and other outdoor activities) inhibit participation.

The provision of culturally and gender sensitive facilities, such as women-only exercise sessions at mosques could serve as a solution for Ontario SA Muslim women to be more active. Studies indicate health promotion programs in religious institutions (e.g. churches) have demonstrated clinical and psychosocial benefit to women of various ethnic groups. Similar to Canadian churches, mosques have key elements identified in the literature to be beneficial in providing physical activity opportunities for Muslim women: partnerships, available and accessible space and supportive social relationships.

To the investigators' knowledge, mosque-based physical activity interventions for SA Muslim women have not been implemented and evaluated in Ontario. Such interventions are needed to help attenuate the risk of diabetes and CHD in this ethnic group who represent a significant part of the Ontario population.

ELIGIBILITY:
Inclusion Criteria:

* Muslim women attending Madinah Mosque

Exclusion Criteria:

men

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of exercise sessions attended | 10 weeks
  Participants are eligible to attend up to 3 exercise sessions per week over a period of 10 weeks. The number of sessions attended will be counted.

SECONDARY OUTCOMES:
Change in Duke Activity Status Index (DASI) | Change from Baseline in DASI at 10 weeks
  The DASI is a self-administered questionnaire that measures functional capacity.

OTHER OUTCOMES:
Change in the International Physical Activity Questionaire (IPAQ) | Change from Baseline in IPAQ at 10 weeks.
  The IPAQ measures health related physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer AD Price, RN,PhD, Principal Investigator — Women's College Hospital; Ananya T Banerjee, RegKin,PhD, Principal Investigator — Women's College Hospital
Locations (1):
- Jennifer Price, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anand SS, Yusuf S, Vuksan V, Devanesen S, Teo KK, Montague PA, Kelemen L, Yi C, Lonn E, Gerstein H, Hegele RA, McQueen M. Differences in risk factors, atherosclerosis, and cardiovascular disease between ethnic groups in Canada: the Study of Health Assessment and Risk in Ethnic groups (SHARE). Lancet. 2000 Jul 22;356(9226):279-84. doi: 10.1016/s0140-6736(00)02502-2. PMID 11071182
- [Background] Chiu M, Austin PC, Manuel DG, Tu JV. Cardiovascular risk factor profiles of recent immigrants vs long-term residents of Ontario: a multi-ethnic study. Can J Cardiol. 2012 Jan-Feb;28(1):20-6. doi: 10.1016/j.cjca.2011.06.002. Epub 2011 Aug 9. PMID 21827964
- [Background] Banerjee AT, Gupta M, Singh N. Patient characteristics, compliance, and exercise outcomes of South Asians enrolled in cardiac rehabilitation. J Cardiopulm Rehabil Prev. 2007 Jul-Aug;27(4):212-8. doi: 10.1097/01.HCR.0000281765.52158.be. PMID 17667016
- [Background] Bryan SN, Tremblay MS, Perez CE, Ardern CI, Katzmarzyk PT. Physical activity and ethnicity: evidence from the Canadian Community Health Survey. Can J Public Health. 2006 Jul-Aug;97(4):271-6. doi: 10.1007/BF03405602. PMID 16967744
- [Background] Williams ED, Stamatakis E, Chandola T, Hamer M. Physical activity behaviour and coronary heart disease mortality among South Asian people in the UK: an observational longitudinal study. Heart. 2011 Apr;97(8):655-9. doi: 10.1136/hrt.2010.201012. Epub 2010 Dec 3. PMID 21131381
- [Background] Carroll R, Ali N, Azam N. Promoting physical activity in South Asian Muslim women through "exercise on prescription". Health Technol Assess. 2002;6(8):1-101. doi: 10.3310/hta6080. No abstract available. PMID 12000689
- [Background] Lawton J, Ahmad N, Hanna L, Douglas M, Hallowell N. 'I can't do any serious exercise': barriers to physical activity amongst people of Pakistani and Indian origin with Type 2 diabetes. Health Educ Res. 2006 Feb;21(1):43-54. doi: 10.1093/her/cyh042. Epub 2005 Jun 13. PMID 15955792
- [Background] Campbell MK, Hudson MA, Resnicow K, Blakeney N, Paxton A, Baskin M. Church-based health promotion interventions: evidence and lessons learned. Annu Rev Public Health. 2007;28:213-34. doi: 10.1146/annurev.publhealth.28.021406.144016. PMID 17155879
- [Background] Banerjee AT, Boyle MH, Anand SS, Strachan PH, Oremus M. The relationship between religious service attendance and coronary heart disease and related risk factors in Saskatchewan, Canada. J Relig Health. 2014 Feb;53(1):141-56. doi: 10.1007/s10943-012-9609-6. PMID 22576676
- [Background] Banerjee AT, Strachan PH, Boyle MH, Anand SS, Oremus M. Attending religious services and its relationship with coronary heart disease and related risk factors in older adults: a qualitative study of church pastors' and parishioners' perspectives. J Relig Health. 2014 Dec;53(6):1770-85. doi: 10.1007/s10943-013-9783-1. PMID 24132458
- [Background] Rolfe DE, Sutton EJ, Landry M, Sternberg L, Price JA. Women's experiences accessing a women-centered cardiac rehabilitation program: a qualitative study. J Cardiovasc Nurs. 2010 Jul-Aug;25(4):332-41. doi: 10.1097/JCN.0b013e3181c83f6b. PMID 20539167
- [Background] Price J, Landry M, Rolfe D, Delos-Reyes F, Groff L, Sternberg L. Women's cardiac rehabilitation: improving access using principles of women's health. Can J Cardiovasc Nurs. 2005;15(3):32-41. PMID 16295796
- [Background] Hlatky MA, Boineau RE, Higginbotham MB, Lee KL, Mark DB, Califf RM, Cobb FR, Pryor DB. A brief self-administered questionnaire to determine functional capacity (the Duke Activity Status Index). Am J Cardiol. 1989 Sep 15;64(10):651-4. doi: 10.1016/0002-9149(89)90496-7. PMID 2782256
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694